CLINICAL TRIAL: NCT01443377
Title: Neoadjuvant Radiochemotherapy Combined With Panitumumab in Locally Advanced KRAS Wild-type Rectal Cancer
Acronym: NEOREC-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-0001021
Record Dates: First submitted 2011-08-23; First posted 2011-09-29 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Rectal Cancer
Keywords: Neorec; rectal cancer; KRAS; Panitumumab; neoadjuvant; Radiochemotherapy; antibody; locally advanced KRAS wild type rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Panitumumab — Intravenous (IV), Panitumumab 6 mg/kg BW q2w d1-d57 (5 times total); begin on day 1 (run-in-phase) and subsequent application on days 15, 29 43 and 57.
  Other Names: Vectibix®

SUMMARY:
This study aims to investigate the combination of panitumumab and a 5-FU-based RCTX in patients with locally advanced KRAS wild-type rectal cancer.

DETAILED DESCRIPTION:
Significant progress in the management of locally advanced rectal cancer has been achieved during the last decade. This includes surgical techniques as the widespread implementation of total mesorectal excision as well as preoperative radiochemotherapy (RCTX). The results of the recent randomized trials led to a current standard in which most (radio-) oncologists now use continuous-infusion 5-FU concomitantly with preoperative radiotherapy. It has been demonstrated that this provides improved tumor downstaging and local control; however, no significant differences have yet been achieved in the 5-year disease-free and overall survival rates.

Thus, the challenge is to integrate more effective systemic therapy into the combined-modality programs. The combination of RCTX with novel chemotherapeutic agents like oxaliplatin and irinotecan in phase I/II trials suggested higher rates of histopathological complete remission (pCR) compared with 5-FU RCTX alone. However, due to the lack of results from randomized trials, to date no improvement of the long-term outcomes could be demonstrated, moreover, for some studies the increased pCR rate was associated with an increase in toxicity.

Another strategy to improve outcome is to incorporate newer, biologically active, targeted therapies into established RCTX regimens. Because of its key role in signalling proliferation, inhibition of apoptosis and angiogenesis the epidermal growth factor receptor (EGFR) is a promising target of antitumor treatment. To date a few clinical phase I/II studies of preoperative RCTX have been initiated to evaluate EGFR inhibitors as radiosensitizer in rectal cancer. These trials demonstrated that a combination of cetuximab and RCTX could be safely applied without dose compromises of the respective treatment components. However, the pCR rates could not be improved in these studies.

Given the strong preclinical rationale to combine EGFR inhibition with RCTX in rectal cancer patients, this study aims to investigate the combination of panitumumab and a 5-FU-based RCTX in patients with locally advanced KRAS wild-type rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, potentially resectable rectal adenocarcinoma staged as uT3/4 N0/1 by endosonography or cT3/4 by MRI of the pelvis with or without local lymph node metastases.
* Wild-type KRAS.
* ECOG-performance status 0 or 1.
* Age ≥ 18 years.
* Laboratory requirements:

  * Haematology: Leucocyte count > 3,000/mm³, neutrophil count ≥1.5x109/L, hemoglobin ≥ 8 g/dL, platelet count ≥100x109/L.
  * Hepatic Function: Total bilirubin ≤ 1.5 time the upper normal limit (UNL), ASAT ≤ 2.5xUNL in absence of liver metastases or ≤ 5xUNL in presence of liver metastases, ALAT ≤ 2.5xUNL in absence of liver metastases or ≤ 5xUNL in presence of liver metastases
  * Renal Function: Creatinine clearance ≥50 mL/min or serum creatinine ≤1.5xUNL
  * Metabolic Function: Magnesium ≥ lower limit of normal, Calcium ≥ lower limit of normal.
* Negative ß-HCG-serum pregnancy test (females of child bearing potential).
* Willing to use double-barrier contraception during study and for 6 months after the end of treatment.
* Ability of patient to understand character and individual consequences of clinical trial
* Written informed consent (must be available before enrollment in the trial)

Exclusion Criteria:

* Prior EGFR targeting or prior chemo- or radiotherapy or tumor surgery.
* Evidence of any distant metastases.
* Manifest or previous secondary malignancies within the last 5 years.
* Uncontrolled infection.
* Clinically significant cardiovascular disease NYHA classification III or IV (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment/randomization.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on screening chest CT scan.
* Diabetes mellitus
* Subject pregnant or breast feeding, or planning to become pregnant within 6 month after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* Active serious illness which renders the patient unsuitable for study entrance, multiple blood sampling or the above mentioned biopsies.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials or observation period of competing trials, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Histopathological complete response rate (pCR) | at week 14 after tumor resection
  pCR determined by means of the resection specimens

SECONDARY OUTCOMES:
Objective tumor response rate assessed by MRI of the pelvis (incl. RECIST) | at day 14 and week 12
Metabolic tumor response rate assessed by means of changes in the standardized uptake values (SUV) using FDG-PET-CT (incl. RECIST) | day 14 and at week 14 before surgery
Pathological tumor regression grades will be classified according to Becker | at week 14 after surgery
Quality of Life (QoL) will be assessed using the EORTC QLQ-C30 in combination with the colorectal cancer-specific quality of life questionaire module (QLQ-CR29) | between day 0 and week 18 end of study
distant metastases-free survival | during follow up every 6 months until death or until 2 years after LPO
  distant metastases-free survival after EOS
relapse-free survival | during follow up every 6 months until death or until 2 years after LPO
  relapse-free survival after end of study
overall survival | during follow up every 6 months until death or until 2 years after LPO
  overall survival after EOS

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jaeger, Prof. Dr, Principal Investigator — National Center of Tumor Disease, Heidelberg
Locations (2):
- Germany (2):
  - National Center for Tumor Disease (NCT), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Nord West, Radioonkologische Klinik, Frankfurt am Main, Hesse